CLINICAL TRIAL: NCT02931292
Title: A Decade of Sleeve Gastrectomy as a Single Bariatric/Metabolic Procedure: Analysis of Short and Long-term Outcome of 562 Patients
Brief Title: A Decade of Sleeve Gastrectomy: Analysis of Short and Long-term Outcome of 562 Patients
Acronym: SG
Status: Completed | Type: Observational
Sponsor: Medical Park Gaziantep Hospital (Other)
Collaborators: Harran University (Other)
Responsible Party: Principal Investigator, Mehmet Kaplan, Principal Investigator, Medical Park Gaziantep Hospital
Other Study IDs: MK-009-MO-SG1
Record Dates: First submitted 2016-10-09; First posted 2016-10-13 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Morbid Obesity; Obesity; Diabetes; Dyslipidemia; Hypertension
Keywords: sleeve gastrectomy; laparoscopy; bariatric surgery; obesity surgery; metabolic surgery
MeSH Terms: conditions — Obesity, Morbid; Obesity; Diabetes Mellitus; Dyslipidemias; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sleeve Gastrectomy: Laparoscopic sleeve gastrectomy
  Interventions: Procedure: Laparoscopic sleeve gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic sleeve gastrectomy — Special care was given to the complete mobilization of the gastric fundus, with meticulous dissection of the posterior gastric wall from the left pillar. A 36-Fr calibration bougie was used. Resection started 2 to 6 cm from pylorus, and it was conducted upward to 1.5 cm from the angle of His, to avoid the "critical area." A gastric remnant of 60-80 mL volume (measured by administering methylene blue saline solution via nasogastric tube) was obtained.

SUMMARY:
Obesity is a chronic disease and its treatment requires close follow-up to accurately assess the efficacy and durability of any treatment strategy. It is widely accepted that bariatric surgery patients require lifetime follow-up to assess for weight loss, co-morbidity changes, and nutritional deficiencies.

The study objective was to ascertain efficacy of weight loss and complication rates in 562 consecutive cases of laparoscopic sleeve gastrectomy (LSG) in a single surgeon practice.

DETAILED DESCRIPTION:
Obesity is a major healthcare problem reaching epidemic proportion and affecting people of all age (1). The only treatment that proven effective option for a significant substantial long-term weight loss and that cures or durably improves comorbidities is still bariatric surgery (2, 3). Because obesity is a chronic disease, it is widely accepted that to accurately assess the efficacy and durability of any type of bariatric surgery requires lifetime follow-up to assess for weight loss, co-morbidity changes, and nutritional deficiencies.

Despite initially performed as a first part of the staged procedures, the laparoscopic sleeve gastrectomy (LSG) has since introduced as a stand-alone bariatric operation associated with good, short and mid-term weight loss and satisfactory complication rates when conducted in experienced hands. Although simplicity and the overall efficacy of the procedure supported by meta-analysis and systematic review (4, 5), there are still limited long-term outcome data (6). Due to publication bias or multiple controversies regarding the technique of LSG, some of the available data may have underreported which has also been resulted in questioning the long-term weight loss efficacy of the procedure.

Although addressed by a recent consensus document,12 there are multiple controversies regarding the technique of LSG, and this may in part be what has led to the variable published results.

The study objective was to assess the long-term (≥ 5 years) as well as short (1 to ≤ 3 years) and mid-term (> 3 to < 5 years) results in regard to the BMI change, resolution of co-morbidities and complications in 562 consecutive morbidly obese patients undergoing LSG as a primary procedure.

ELIGIBILITY:
Inclusion Criteria:

* underwent LSG for morbid obesity and related morbidities as a primary procedure

Exclusion Criteria:

* previous history of obesity surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From Jun 2005 to Jun 2015, overall 562 consecutive morbidly obese patients admitted to the Hatem Hospital and Medical park Gaziantep Hospital that underwent sleeve gastrectomy for morbid obesity and/or its related co-morbidities were included to the study.
Sampling Method: Probability Sample
Enrollment: 562 (Actual)
Dates: Start 2005-06; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Percent excess body mass index loss (%EBMIL) | through study completion, an average of 1 year
  calculated using formula: %EBMIL = [∆BMI / (initial BMI - 25)] x 100

SECONDARY OUTCOMES:
Hemoglobin A1c (HbA1c) | through study completion, an average of 1 year
  Definitions of glycemic outcomes after sleeve gastrectomy
change on lipid profile | through study completion, an average of 1 year
  Change on lipid profile before and after bariatric surgery was reported according to the Adult Treatment Panel III Guidelines, 2001, of the National Heart, Lung and Blood Institute as follows: no change, improvement in dislipidemia (defined as decrease in number or dose of lipid-lowering agents with equivalent control of dyslipidemia or improved control of lipids on equivalent medication) and remission (defined as normal lipid panel off medication).
percent of complications | through study completion, an average of 1 year
  Complications were evaluated under two headings. Major complications were defined as any complication that resulted in a prolonged hospital stay (beyond 7 days), reintervention, or reoperation. Minor complications were included everything else that is not included under major. They were further categorized as early if observed in 30 days or late if beyond 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Kaplan, M.D., Principal Investigator — Bahcesehir University, BAU

IPD SHARING:
Plan to Share IPD: No